CLINICAL TRIAL: NCT00503776
Title: Randomized Pilot Trial of Chemoradiation Plus or Minus Amifostine to Assess Potential Nutritional, Inflammatory and Physical Outcomes Related to Xerostomia, Mucositis and Dysphagia
Brief Title: Chemo/XRT +/- Amifostine to Assess Outcomes Related to Xerostomia, Mucositis, & Dysphagia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding became unavailable
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine; Director, Cancer Supportive Care Program; Director, Head and Neck Research Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC HN 0554; VU-VICC-HN-0554; VU-VICC-IRB-051068
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Dysphagia; Head and Neck Cancer; Mucositis; Xerostomia
Keywords: xerostomia; mucositis; dysphagia; radiation toxicity; chemotherapeutic agent toxicity; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; salivary gland squamous cell carcinoma; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer
MeSH Terms: conditions — Deglutition Disorders; Head and Neck Neoplasms; Mucositis; Xerostomia; Radiation Injuries; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Amifostine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm IA (Active Comparator): Patients undergo specialized nutrition therapy (SNT) including dietitian counseling and calorie goal instruction.
  Interventions: Procedure: therapeutic dietary intervention
- Arm IB (Active Comparator): Patients undergo SNT and low weight resistance training (LWRT).
  Interventions: Behavioral: exercise intervention; Procedure: therapeutic dietary intervention
- Arm IIA (Experimental): Patients receive amifostine subcutaneously (SC) 30-60 minutes prior to each dose of intensity-modulated radiotherapy (IMRT). Patients also undergo SNT as in arm IA.
  Interventions: Drug: amifostine trihydrate; Procedure: therapeutic dietary intervention
- Arm IIB (Experimental): Patients receive amifostine SC 30-60 minutes prior to each dose of IMRT. Patients also undergo SNT and LWRT as in arm IB.
  Interventions: Behavioral: exercise intervention; Drug: amifostine trihydrate; Procedure: therapeutic dietary intervention

INTERVENTIONS:
Behavioral: exercise intervention — Patients undergo low weight resistance training.
  Arms: Arm IB; Arm IIB
Drug: amifostine trihydrate — Given subcutaneously
  Other Names: Ethyol
  Arms: Arm IIA; Arm IIB
Procedure: therapeutic dietary intervention — Patients undergo specialized nutrition therapy (SNT) including dietitian counseling and calorie goal instruction.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Amifostine may decrease the side effects caused by chemotherapy and radiation therapy. It is not yet known whether chemotherapy and radiation therapy are more effective with or without amifostine in treating head and neck cancer.

PURPOSE: This randomized phase II trial is studying amifostine to see how well it works compared with standard care in reducing side effects in patients undergoing chemotherapy and radiation therapy for stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the incidence and severity of acute and chronic swallowing dysfunction in stage III or IV head and neck cancer patients receiving concurrent chemoradiation with or without amifostine

Secondary

* To assess the relative incidence and severity of acute and chronic xerostomia in stage III or IV head and neck cancer patients receiving chemoradiation with or without amifostine.
* To assess the relative incidence and severity of mucositis and mucositis-related inflammation in stage III or IV head and neck cancer patients receiving chemoradiation with or without amifostine.
* To assess the effects of dysphagia, xerostomia, and mucositis-related inflammation on nutritional, physical, and functional status

OUTLINE: Patients undergo intensity-modulated radiotherapy (IMRT) and concurrent chemotherapy comprising carboplatin and paclitaxel weekly.

Patients are randomized to 1 of 2 treatment arms.

* Arm I (standard of care): Patients are further divided into 1A or 1B.

  * Arm IA: Standard of care plus standardized nutrition therapy (SNT)
  * Arm IB: Standard of care plus standardized nutrition therapy plus low weight resistance training (LWRT).
* Arm II (amifostine): Patients are further divided into 2A or 2B.

  * Arm IIA: Amifostine 500mg diluted in 2.9 ml injected 30-60 minutes prior to each radiation dose plus standardized nutrition therapy
  * Arm IIB: Amifostine 500mg diluted in 2.9 ml injected 30-60 minutes prior to each radiation dose plus standardized nutrition therapy plus low weight resistance training

In all arms, patients undergo swallowing function, dietary, body composition, muscle, and physical and functional performance measurements at baseline and at 1, 3, and 6 months post-therapy. Quality of life, salivary production, fatigue, and symptoms (including swallowing/eating foods, appetite, weight loss/nutrition, pain, and speech/communication) are assessed at baseline and at 1, 3, and 6 months post-therapy. Anthropometric measurements are also performed at the above time points and at mid-therapy.

Blood samples and buccal rinses are collected at baseline and at 1, 3, and 6 months post-therapy for biomarker studies and for proteomic and genomic analysis by liquid chromatography and tandem mass spectrometry.

After completion of study treatment, patients are followed at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria

* Age greater than 21
* Biopsy proven stage 3 or 4 squamous cell carcinoma of the larynx, pharynx, oral cavity or salivary glands
* No prior history of active cancer within three years other than non-melanoma skin cancer, early stage prostate or early stage cervical cancer
* controlled co-morbid disease
* ECOG PS of 0-3
* Plan for definitive or post-operative CCR within 4 weeks
* Written informed consent
* Working telephone
* May have received prior induction chemotherapy
* Agree to use only study supplied liquid nutrition supplements or dietary supplements, for per os or feeding tube intake

Exclusion Criteria

* Diagnosed HIV or AIDS
* History of ETOH or drug abuse within 3 months
* Pregnant or lactating
* On steroid medication or prescribed NSAIDs
* Consuming specialty nutrition supplements containing additional amounts of eicosapentaenoic acid (EPA) or docosahexaenoic acid (DHA)
* On orexigenic (appetite stimulant) medication.
* Uncontrolled comorbid disease defined as: a) severe cardiac disease Class III or greater; b) blood pressure > 160/95; c) uncontrolled pain
* Does not have working telephone.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to accrual from 01/01/2006 through 03/05/2008.
Pre-assignment Details: 43 patients consented, one was ineligible for a total of 42 patients on study.
Period: Overall Study
Arm/Group | Arm IA | Arm IB | Arm IIA | Arm IIB
Started | 8 | 12 | 12 (one patient withdrew before receiving protocol therapy) | 10 (one patient withdrew before receiving protocol therapy)
Completed | 7 | 12 | 10 | 8
Not Completed | 1 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm IA | Arm IB | Arm IIA | Arm IIB | Total
Number analyzed (Participants) | 8 | 12 | 12 | 10 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 10 | 10 | 40
  >=65 years | 0 | 0 | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (1) | 55 (1) | 54 (1) | 55 (1) | 54 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 0 | 6
  Male | 5 | 11 | 10 | 10 | 36
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 12 | 10 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Each Degree of Swallowing Dysfunction
Description: Grade of swallowing dysfunction as measured by the modified barium swallow score: grade 1, normal; grade 2, within functional limits; grade 3, mild impairment; grade 4, mild to moderate impairment; grade 5, moderate impairment; grade 6, moderate to severe impairment; grade 7, severe impairment
Time Frame: 6 months after concurrent chemotherapy and radiation
Population: One patient (Arm 2B) did not undergo the 6-month study
Measure: Number; unit: participants
Groups:
- Arm IB: Patients undergo SNT and low-weight resistance training (LWRT).
Arm/Group | Arm IA | Arm IB | Arm IIA | Arm IIB
Number analyzed (Participants) | 8 | 12 | 12 | 9
participants
  No. of patients with dysphagia grade 0 | 2 | 1 | 2 | 3
  No. of patients with dysphagia grade 1 | 1 | 5 | 4 | 4
  No. of patients with dysphagia grade 2 | 1 | 1 | 2 | 1
  No. of patients with dysphagia grade 3 | 3 | 1 | 1 | 0
  No. of patients with dysphagia grade 4 | 0 | 0 | 0 | 0
  Not Accessible | 1 | 4 | 3 | 1

2. Secondary Outcome: Stimulated and Unstimulated Salivary Production
Description: Unstimulated and stimulated salivary production, measured in mL/minute. Unstimulated salivary production is determined by expectoration of passively accumulated secretions accumulated in three 2-minute periods. Stimulated salivary production is determined by chewing paraffin wax with expectoration of passively accumulated secretions accumulated in three 2-minute periods.
Time Frame: 6 months after concurrent chemotherapy and radiation
Population: Patients who underwent salivary testing at 6 months. The following patients were not available at 6- months for testing for salivary production: Arm 1A (1), Arm 1B (4), Arm 2A (3), Arm 2B (2)
Measure: Mean (Standard Deviation); unit: mL per minute
Arm/Group | Arm IA | Arm IB | Arm IIA | Arm IIB
Number analyzed (Participants) | 7 | 8 | 9 | 8
mL per minute
  Unstimulated | 0.64 (0.37) | 1.70 (1.44) | 1.38 (1.90) | 0.68 (0.32)
  Stimulated | 0.72 (1.85) | 5.04 (3.16) | 5.25 (3.39) | 0.94 (2.25)

3. Secondary Outcome: Number of Patients With Oral Mucositis by Grade
Description: Measured by Common Toxicity Criteria (CTC) v. 3.00 = no mucositis (minimum score), 1 = mild mucositis, 2 = moderate mucositis, 3 = severe mucositis, 4 = life-threatening, disabling mucositis, 5 = death (worst score).
Time Frame: 6 months after concurrent chemotherapy and radiation
Population: Participants available for 6-month follow-up oral examination. No 6-month follow-up data were available for the following numbers of patients: Arm 1A (1), Arm 1B (4), Arm 2A (3), Arm 2B (2).
Measure: Number; unit: participants
Arm/Group | Arm IA | Arm IB | Arm IIA | Arm IIB
Number analyzed (Participants) | 7 | 8 | 9 | 8
participants
  No. of patients with grade 0, no mucositis | 3 | 4 | 6 | 3
  No. of patients with grade 1, mild mucositis | 0 | 4 | 2 | 3
  No of patients with grade 2, moderate mucositis | 1 | 0 | 1 | 2
  No of patients with grade 3, severe mucositis | 3 | 0 | 0 | 0
  No. of patients with grade 4, disabling mucositis | 0 | 0 | 0 | 0
  No. of patients with grade 5 mucositis, death | 0 | 0 | 0 | 0

4. Secondary Outcome: Changes in the Amount and Texture of Food Consumed
Description: Patients are asked to note their food intake in terms of amount and texture over the past 24 hours as measured by 24-hour dietary recalls.
Time Frame: at baseline, at 1 month, 3 months and 6 months post-chemoradiation
Population: Due to loss of funding, sufficient data for analysis was not collected.
Arm/Group | Arm IA | Arm IB | Arm IIA | Arm IIB
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Changes in the Frequency and Types of Dietary Intakes
Description: Patients are asked to note their food intake in terms of amount and texture over the past 24 hours as measured by 24 hour dietary recalls.
Time Frame: at baseline, at 1 month, 3 months and 6 months post-chemoradiation
Population: Due to loss of funding, sufficient data for analysis was not collected.
Arm/Group | Arm IA | Arm IB | Arm IIA | Arm IIB
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm IA | Arm IB | Arm IIA | Arm IIB
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/12 | 2/12 | 4/9
Other Adverse Events (participants affected / at risk) | 7/8 | 12/12 | 10/12 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm IA (N=8) | Arm IB (N=12) | Arm IIA (N=12) | Arm IIB (N=9)
accute hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
mucositis/stomatitis-oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Muscle weakness - lower extremity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - abdomen NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pain - larynx (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
pain - oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pain - NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pain - rectal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever-in absence of neutropenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rigor, chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils-blood (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
edema limb (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm IA (N=8) | Arm IB (N=12) | Arm IIA (N=12) | Arm IIB (N=9)
constipation (Gastrointestinal disorders) | 7 (22) | 10 (23) | 9 (24) | 6 (14)
diarrhea (Gastrointestinal disorders) | 4 (8) | 3 (4) | 3 (4) | 3 (4)
difficulty chewing (Gastrointestinal disorders) | 6 (17) | 11 (30) | 9 (29) | 8 (23)
dysphagia (Gastrointestinal disorders) | 7 (32) | 12 (46) | 10 (42) | 8 (34)
mucositis (Gastrointestinal disorders) | 7 (29) | 12 (40) | 9 (33) | 8 (32)
nausea (Gastrointestinal disorders) | 7 (21) | 6 (13) | 8 (17) | 8 (15)
vomiting (Gastrointestinal disorders) | 6 (13) | 6 (12) | 8 (12) | 6 (8)
dry mouth (Gastrointestinal disorders) | 7 (32) | 12 (46) | 10 (40) | 8 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes